CLINICAL TRIAL: NCT02988219
Title: Evaluation of Cardiac Arrhythmias in Patients Undergoing Kidney Cancer Surgery Depending on the Anaesthesia Method
Brief Title: Cardiac Arrhythmias in Patients Undergoing Kidney Cancer Surgery Depending on the Anaesthesia Method
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Karolina Dobrońska, M.D., Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: U/1/2010
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Arrhythmia, Cardiac; Kidney Cancer; Surgery; Anesthesia, Local
Keywords: cardiac arrhythmia; epidural anesthesia; combined anesthesia; general anesthesia; NSS; radical nephrectomy; extraperitoneal
MeSH Terms: conditions — Arrhythmias, Cardiac; Kidney Neoplasms | interventions — Bupivacaine; Fentanyl; Anesthesia, General; Intubation; Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia (G) (Active Comparator): Holter ECG monitor General anesthesia Open kidney cancer surgery
  Interventions: Device: Holter ECG monitor; Procedure: Open kidney cancer surgery; Procedure: General anesthesia
- Combined general/epidural (G/E) (Experimental): Holter ECG monitor Epidural anesthesia General anesthesia Open kidney cancer surgery
  Interventions: Drug: Bupivacaine-fentanyl; Device: Holter ECG monitor; Procedure: Open kidney cancer surgery; Procedure: General anesthesia; Procedure: Epidural Anaesthesia

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — Local anesthetic
  Other Names: Marcaine; Sensorcaine; Astra Zeneca; Bupivacaine-epinephrine; Fentanyl
  Arms: Combined general/epidural (G/E)
Device: Holter ECG monitor — 3-chanel, CM5 leads
Procedure: Open kidney cancer surgery — Lateral position
  Other Names: nephron sparing surgery (NSS); Radical nephrectomy; Extraperitoneal
Procedure: General anesthesia
  Other Names: Intubation; Fentanyl; Narcosis
Procedure: Epidural Anaesthesia
  Other Names: Bupivacaine; Epidural catheter
  Arms: Combined general/epidural (G/E)

SUMMARY:
This study evaluates the incidence of cardiac arrhythmias during the perioperative period in patients undergoing open kidney cancer surgery in the lateral position. All the participants will be randomly allocated to receive general (Group G) or combined epidural/general anaesthesia (Group G/E). The anaesthetic technique is standardized. The Holter monitor will be applied at the evening before the surgery, tracing continuously for a period of 24 hours (7PM-7PM)

DETAILED DESCRIPTION:
Cardiac arrhythmias are a common complication during and after cardio-thoracic surgery. They are also a major source of morbidity and mortality. After general surgery, they usually do not require clinically significant management but the literature on this topic is obsolete. There is no literature data about their incidence during kidney surgery in the lateral position when the bed is scissored so the legs and head are low. The aim of this study was to define what types of arrhythmias are the most common during kidney cancer surgery, their incidence and whether combining general with epidural anesthesia prevents them.

An approval from the Medical University of Warsaw Bioethical Committee has been obtained. Patients need to give written informed consent to participate in the study.

It is anticipated that 50 patients with open kidney cancer surgery performed in the lateral position, under general or combined anesthesia will be enrolled.

A Holter ECG monitor (3-chanel, leads CM5) will be applied at the evening before the surgery, tracing continuously for a period of 24 hours (7PM-7PM).

Patients will be randomly allocated (random permuted blocks within strata) to receive general or combined epidural/general anesthesia. The anesthetic technique is standardized. All the data registered by the Holter ECG monitor will be analyzed and compared with the nursery and anesthesia records.

ELIGIBILITY:
Inclusion Criteria:

* Open renal cell carcinoma surgery, lateral position
* American Society of Anesthesiologists (ASA) physical grade I-III
* No history of cardiac arrhythmias
* Informed consent

Exclusion Criteria:

* Pregnancy and breast feeding
* Contraindications for epidural anesthesia
* Laparoscopic or robotic surgery
* Suspected difficult intubation (ex. fibroscopic)
* Chest deformations
* Prior cardiac/thoracic surgery
* Cardiac insufficiency
* abnormal ECG before the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Dobronska, MD, Principal Investigator — I Department of Anaesthesiology and Intensive Care
Locations (1):
- I Department of Anaesthesiology and Intensive Care, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dobronska K, Jureczko L, Kowalczyk R, Dobronski P, Trzebicki J. Open kidney cancer surgery and perioperative cardiac arrhythmias. Cent European J Urol. 2020;73(4):432-439. doi: 10.5173/ceju.2020.1734. Epub 2020 Nov 2. PMID 33552568

RESULTS

PARTICIPANT FLOW:
Groups:
- General Anesthesia (G): General anesthesia Holter ECG monitor: 3-chanel, CM5 leads Open kidney cancer surgery: Lateral position
- Combined General/Epidural (G/E): General anesthesia Epidural anesthesia: Local anesthetic Holter ECG monitor: 3-chanel, CM5 leads Open kidney cancer surgery: Lateral position
Period: Overall Study
Arm/Group | General Anesthesia (G) | Combined General/Epidural (G/E)
Started | 25 | 25
Completed | 24 | 22
Not Completed | 1 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia (G) | Combined General/Epidural (G/E) | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 7 | 2 | 9
Age, Continuous [Median (Standard Deviation); unit: years] | 61 (8.50) | 57 (9.04) | 59 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  Poland | 24 | 22 | 46
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 28.14 (4.84) | 30.04 (7.01) | 29.29 (5.99)
ASA [Median (Full Range); unit: scores on a scale] — AMERICAN SOCIETY OF ANESTHESIOLOGISTASA (ASA) PHYSICAL STATUS CLASSIFICATION SYSTEM
  ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  *The addition of "E" denotes Emergency surgery
  scores on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Type of Surgery [Count of Participants; unit: Participants]
  NSS | 12 | 17 | 29
  Nefrectomy | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Perioperative Cardiac Arrhythmias Evaluated by a Continuous ECG Holter Monitoring in the Perioperative Period
Description: The investigator evaluates the incidence of cardiac arrhythmias, the type of arrhythmias and whether additional interventions were needed to treat them
  Arrhythmias observed:
  tachycardia >100 bpm bradycardia < 50 bpm pause (P-P interval > 2 seconds) ventricular extrasystoles (VE) > 1000/ 24 hours supraventricular extrasystoles (SVE) >200/24 hours
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Groups:
- Combined General/Epidural (G/E): General anesthesia Epidural anesthesia: Local anesthetic Holter ECG monitor: 3-chanel, CM5 leads Open kidney cancer surgery: Lateral position General anesthesia
Arm/Group | General Anesthesia (G) | Combined General/Epidural (G/E)
Number analyzed (Participants) | 24 | 22
Participants
  Tachycardia < 140 bpm before surgery: observed | 6 | 6
  Tachycardia < 140 bpm before surgery: not observed | 18 | 16
  Tachycardia < 140 bpm during surgery: observed | 2 | 5
  Tachycardia < 140 bpm during surgery: not observed | 22 | 17
  Tachycardia < 140 bpm after surgery: observed | 5 | 4
  Tachycardia < 140 bpm after surgery: not observed | 19 | 18
  Bradycardia before surgery: observed | 3 | 3
  Bradycardia before surgery: not observed | 21 | 19
  Bradycardia during surgery: observed | 14 | 10
  Bradycardia during surgery: not observed | 10 | 12
  Bradycardia after surgery: observed | 6 | 4
  Bradycardia after surgery: not observed | 18 | 18
  Bradycardia in the perioperative period: observed | 16 | 11
  Bradycardia in the perioperative period: not observed | 8 | 11
  pause > 2s before surgery: observed | 0 | 0
  pause > 2s before surgery: not observed | 24 | 22
  pause > 2s during surgery: observed | 2 | 0
  pause > 2s during surgery: not observed | 22 | 22
  pause > 2s after surgery: observed | 2 | 2
  pause > 2s after surgery: not observed | 22 | 20
  pause > 2s in the perioperative period: observed | 2 | 2
  pause > 2s in the perioperative period: not observed | 22 | 20
  SVE before surgery: observed | 1 | 0
  SVE before surgery: not observed | 23 | 22
  SVE during surgery: observed | 1 | 1
  SVE during surgery: not observed | 23 | 21
  SVE after surgery: observed | 1 | 2
  SVE after surgery: not observed | 23 | 20
  SVE in the perioperativ: observed | 1 | 2
  SVE in the perioperativ: not observed | 23 | 20
  VE before surgery: observed | 1 | 1
  VE before surgery: not observed | 23 | 21
  VE during surgery: observed | 3 | 1
  VE during surgery: not observed | 21 | 21
  VE after surgery: observed | 3 | 2
  VE after surgery: not observed | 21 | 20
  VE in the perioperative period: observed | 3 | 3
  VE in the perioperative period: not observed | 21 | 19
  Additional intervention needed: observed | 0 | 0
  Additional intervention needed: not observed | 24 | 22
Statistical Analysis 1: Comparison: General Anesthesia (G) vs Combined General/Epidural (G/E); Bradycardia during surgery; Test type: Superiority or Other; p = 0.3861, Chi-squared
Statistical Analysis 2: Comparison: General Anesthesia (G) vs Combined General/Epidural (G/E); No bradycardia observed in the perioperative period; Test type: Superiority or Other; p = 0.2591, Chi-squared

2. Secondary Outcome: The Prevention of Cardiac Arrhythmias Occurence by Epidural Anesthesia Added to General Anesthesia Evaluated by a Number and Type of Arrhythmias Observed
Description: The investigator evaluates the incidence of cardiac arrhythmias depending on anesthesia method by observing the number and type of arrhythmias and whether additional interventions were needed to treat them
Time Frame: 60 months
Population: arrhythmias analysed: bradycardia, pause > 2s, supraventricular extrasystoles, ventricular extrasystoles; corrected QT interval (QTc)
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia (G) | Combined General/Epidural (G/E)
Number analyzed (Participants) | 24 | 22
Participants
  arrhythmia before surgery: observed | 3 | 4
  arrhythmia before surgery: not observed | 21 | 18
  arrhythmia during surgery: observed | 16 | 12
  arrhythmia during surgery: not observed | 8 | 10
  arrhythmia after surgery: observed | 8 | 6
  arrhythmia after surgery: not observed | 16 | 16
  QTc long > 0.45s before surgery: observed | 0 | 0
  QTc long > 0.45s before surgery: not observed | 24 | 22
  QTc long > 0.45s during surgery: observed | 0 | 2
  QTc long > 0.45s during surgery: not observed | 24 | 20
  QTc long > 0.45s after surgery: observed | 1 | 6
  QTc long > 0.45s after surgery: not observed | 23 | 16
  QTc long > 0.45s in the perioperative time: observed | 1 | 8
  QTc long > 0.45s in the perioperative time: not observed | 23 | 14
  Additional intervention needed: observed | 0 | 0
  Additional intervention needed: not observed | 24 | 22
Statistical Analysis 1: Comparison: General Anesthesia (G) vs Combined General/Epidural (G/E); Arrhythmia before surgery; Test type: Superiority or Other; p = 0.597, Chi-squared
Statistical Analysis 2: Comparison: General Anesthesia (G) vs Combined General/Epidural (G/E); arrhythmia during surgery; Test type: Superiority or Other; p = 0.4, Chi-squared
Statistical Analysis 3: Comparison: General Anesthesia (G) vs Combined General/Epidural (G/E); arrhythmia after surgery; Test type: Superiority or Other; p = 0.6544, Chi-squared
Statistical Analysis 4: Comparison: General Anesthesia (G) vs Combined General/Epidural (G/E); long QTc > 0.45s after surgery; Test type: Superiority or Other; p = 0.077, Chi-squared
Statistical Analysis 5: Comparison: General Anesthesia (G) vs Combined General/Epidural (G/E); long QTc > 0.24 s in the perioperative time; Test type: Superiority or Other; p = 0.0174, Chi-squared

ADVERSE EVENTS:
Arm/Group | General Anesthesia (G) | Combined General/Epidural (G/E)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes